CLINICAL TRIAL: NCT06883058
Title: Implementation of the Caregivers-Patients Support Coping with Advanced-Cancer (CASA) Intervention.
Acronym: CASA pre-pilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ponce Medical School Foundation, Inc. (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2411224820
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Advanced Cancer; Caregivers; Patients; Stage III Cancer; Stage IV Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Placebo Comparator): Usual care will be provided to participants in the control group. The usual care consists of symptom management once a week and 5 sessions.
  Interventions: Behavioral: Placebo
- CASA (Experimental): The Caregivers-Patients Support Intervention for Advanced Cancer (CASA) will be delivered to patients and caregivers. The sessions follow a protocol and will be held weekly or bi-weekly for a total of 5 sessions.
  Interventions: Behavioral: Caregivers-patients support intervention for advanced cancer (CASA)

INTERVENTIONS:
Behavioral: Caregivers-patients support intervention for advanced cancer (CASA) — The Caregivers-Patients Support Intervention for Advanced Cancer (CASA) will be delivered to patients and caregivers. The sessions follow a protocol and will be held weekly or bi-weekly for a total of 5 sessions.
  Arms: CASA
Behavioral: Placebo — Usual care will be provided to participants in the control group. The usual care consists of symptom management once a week and 5 sessions.
  Arms: Usual Care

SUMMARY:
This pre-pilot aims to prepare the PI to receive hands-on experience in implementation and dissemination and design and lead pilot studies in palliative care. The catchment area communities experience lower cancer health outcomes and are more likely to be diagnosed with advanced cancer when compared to other surrounding areas. The PI's catchment area experiences advanced cancer, and their caregivers are at an increased risk for unmet psychosocial needs; this pre-pilot will allow the PI to focus on this critical gap in equal healthcare. The research goal of this proposal is to refine and pre-pilot an intervention titled Caregivers Patients Support to Cope with Advanced Cancer (CASA), a five-session, 60-minute telehealth series for patient-caregiver dyads. The rationale for this project is that it will lay the groundwork for a Randomized Control Trial (RCT) testing the efficacy of CASA. It will also assess the implementation of an innovative method to deliver the CASA intervention. This study aims to use the collaborative intervention planning framework and ORBIT model to modify and assess the feasibility and preliminary effect of the CASA intervention. The overall impact of this study is to improve access to psychosocial, culturally adapted interventions in the proposed catchment area.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients must be stage III and IV solid tumor patients who report distress >4 on the Distress Thermometer
* Caregivers. Identified caregivers by distressed patients.

Exclusion Criteria:

* (1) diagnosed with a major disabling medical or psychiatric condition, (2) unable to understand the consent procedure, or (3) too ill to participate, all as reported by the participant and/or determined by the investigator's judgment.

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-12 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
FACIT-Sp | 5 minutes
  is a 12-item questionnaire that measures spiritual well-being in people with cancer and other chronic illnesses. Cancer patients, psychotherapists, and religious/spiritual experts provided input on the development of the items.

SECONDARY OUTCOMES:
PHQ-9 | 5 minutes
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression.
GAD-7 | 5 minutes
  The Generalized Anxiety Disorder 7-item (GAD-7) is a easy to perform initial screening tool for generalized anxiety disorder

IPD SHARING:
Plan to Share IPD: Undecided